CLINICAL TRIAL: NCT06450288
Title: Effectiveness of the Green Oasis (GO) Wellness Program for Residents Living in Concordia Tsat Sing Kong Transitional Housing Estate
Brief Title: Effectiveness of GO for Transitional Housing Residents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GO
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Quality of Life; Wellness, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GO group (Experimental): Participants who reside in the Concordia Tsat Sing Kong Transitional Housing Estate (still under construction) will be invited to join the GO wellness program.
  Interventions: Behavioral: GO

INTERVENTIONS:
Behavioral: GO — Green Oasis wellness program: include physical exercises, gardening, interaction with the developed website. Participants' general health status and website evaluation will be measured at T0 (baseline), T1 (3 months), T2 (9 months), using standardized questionnaires.
  Study Design: pre-post study, 50 participants will be recruited from the Concordia Tsat Sing Kong transitional housing estate.

SUMMARY:
The goal of this pre-post study is to enhance the health and wellness of the residents in the Concordia Tsat Sing Kong Transitional Housing Estate. This study aims to evaluate the effectiveness of the Green Oasis (GO) wellness program in:

1. Increase health awareness and engaging in health promoting activities, including more physical activities/walking, gardening.
2. Enhance happiness and quality of life.

Participants will:

* complete physical exercises, gardening, and interact with the GO website
* receive health talks

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 or above.
* Scored >6 in the Abbreviated Mental Test; a cut-off point of 6 is valid in differentiating between normal and abnormal cognitive functions for geriatric clients.
* Can understand Cantonese.
* Able to take part in light exercise and stretching.
* Have access to smartphone and internet.

Exclusion Criteria:

* Have a serious organic disease or malignant tumor.
* Have a mental disorder diagnosed by neurologists or psychiatrists.
* Experienced drug addiction

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (World Health Organization) | T0 (baseline), T1 (6 months), T2 (12 months)
  Conducting pre- and post-test of WHOQOL-BREF. The brief, Chinese version of the World Health Organization's quality of life scale (WHOQOL-BREF) has our domains: physical health, psychological health, social relationships, and environment. A 5-point response scale is used in the scale. Higher scores indicate higher quality of life. WHOQOL-BREF has good validity and reliability.
Happiness | T0 (baseline), T1 (6 months), T2 (12 months)
  Conducting pre- and post-test of Subjective Happiness Scale (SHS). The Subjective Happiness Scale's Chinese adaptation (SHS) consists of 4 items to measure individual levels of subjective happiness. It features 4 questions, each evaluated on a 7-point Likert scale, where a higher score signifies a higher degree of subjective happiness
Activities of daily living | T0 (baseline), T1 (6 months), T2 (12 months)
  Conducting pre- and post-test of Activities of Daily Living Questionnaire (ADLQ). The activities of daily living questionnaire (ADLQ) will be measured by the Barthel Index, which consists of 10 items of ADL, including mobility and self-care ability. It refers to the basic self-care tasks that individuals perform daily to maintain their overall well-being and take care of themselves; the activities include eating, grooming, bathing, and dressing.
Physical activity | T0 (baseline), T1 (6 months), T2 (12 months)
  Conducting pre- and post-test of the 5-Item Physical Activity Questionnaire. The Chinese adoption of the 5-item physical activity questionnaire will be used to assess the physical activity levels of the participants. This questionnaire uses a 5-point Likert scale to assess five items: frequency, duration, intensity, overall length, and type of activities the participants perform during their spare times. The test-retest reliability of this questionnaire is between 0.61 and 0.91, indicating its usefulness.
Satisfaction with migration life | T0 (baseline), T1 (6 months), T2 (12 months)
  Conducting pre- and post-test of the Satisfaction With Migration Life Scale (SWMLS). The Chinese adoption of the Satisfaction With Migration Life Scale (SWMLS) to assess participants' satisfaction with their life after moving in to transitional housing. The scale has 5 questions in total and follows a 7-point Likert scale, with some modifications on the wordings according to the study. SWMLS has good validity and reliability.
Pain intensity | T0 (baseline), T1 (6 months), T2 (12 months)
  Pain will be measured using the Chinese version of the Brief Pain Inventory to assess the multidimensional nature of the participants' pain, including intensity and interference with daily activities over the past 24 hours. The total scores for pain severity (four items) range from 0 to 10, with higher scores indicating more severe pain. This scale demonstrated good reliability, with coefficient alphas greater than 0.70

SECONDARY OUTCOMES:
Website evaluation | 2 weeks after T2 (post-test)
  Website will be assessed using the Chinese version of the System Usability Scale (SUS). The SUS consists of 10 items rated using a 5-point Likert scale. A higher total score indicates better quality of the rated system. This scale has good reliability, with a Cronbach's alpha of 0.84.
Semi-structured interview | within 2 weeks after T2 (post-test)
  Interview participants about joining the program, their perceived benefits, challenges, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong